CLINICAL TRIAL: NCT02630524
Title: Diet Composition and Cardiometabolic Risk Reduction in Adults With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Brooks C. Wingo, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F151001005
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Obesity; Spinal Cord Injuries; Diabetes
MeSH Terms: conditions — Obesity; Spinal Cord Injuries; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Carbohydrate Diet (Experimental)
  Interventions: Behavioral: eHealth Behavioral Lifestyle Intervention Device: Telecoach
- Standard Diet (Active Comparator)
  Interventions: Behavioral: eHealth Behavioral Lifestyle Intervention Device: Telecoach

INTERVENTIONS:
Behavioral: eHealth Behavioral Lifestyle Intervention Device: Telecoach — Participants will receive weekly/biweekly coaching sessions with a telecoach and use eHealth platform to log food and exercise, review daily goals, and find strategies for reaching goals.

SUMMARY:
The purpose of this study is to examine the effectiveness of a low carbohydrate diet on increasing dietary adherence and improving cardiometabolic risk factors among adults with spinal cord injury (SCI). Seventy overweight/obese adults with SCI will be randomized to one of two groups: 1) a reduced carbohydrate diet or 2): a "standard" diet (STD). Participants will take part in a 6-month behavioral lifestyle intervention implemented through a novel eHealth platform specially designed for individuals with SCI.

ELIGIBILITY:
Inclusion Criteria:

* SCI ≥ 1 year post injury
* able to use arms for exercise
* BMI of 22-50 kg/m2
* 19-60 years old
* reliable access to internet and smartphone
* have the ability to converse in English
* ability to prepare own food or have input into person responsible for food preparation

Exclusion Criteria:

* heart disease
* renal disease
* active pressure sore
* persons on medically restricted diets

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Adherence to prescribed macronutrient composition as measured by multiple pass 24 hour dietary recall | 6 months
  Participants will record 3 days of food intake at each measurement time point. Calories and macronutrient values from the 3 days will be averaged. We will calculate an adherence score using methodology described by Alhassan et al. Adherence will be measured as the difference between recorded intake and prescribed intake of the macronutrient of interest for each group (i.e., carbohydrates for the low carbohydrate group, fat for the standard group). For example, if a participant in the low carbohydrate group is prescribed a limit of 50g of CHO/day, and recorded intake is 70g, the adherence score will be 20. A score of 0 indicates meeting recommended values, and higher scores indicate poorer adherence than lower scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeshore Foundation, Birmingham, Alabama, United States